CLINICAL TRIAL: NCT04423991
Title: Identification of a Responsive Subpopulation to Hydroxychloroquine in COVID-19 Patients Using Machine Learning: the IDENTIFY Trial
Brief Title: Identification of a Responsive Subpopulation to Hydroxychloroquine in COVID-19 Patients Using Machine Learning
Acronym: IDENTIFY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dascena (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 060820
Record Dates: First submitted 2020-06-08; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: COVID-19; Coronavirus; Mortality
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exposed group (Experimental): All patients were exposed to the algorithm and were characterized as being likely responders to hydroxychloroquine treatment. Treatment decisions regarding the administration of hydroxychloroquine were made independently by care providers.
  Interventions: Device: COViage

INTERVENTIONS:
Device: COViage — Machine learning intervention

SUMMARY:
The purpose of this study was to assess the performance of a machine learning algorithm which identifies patients for whom hydroxychloroquine treatment is associated with predicted survival.

DETAILED DESCRIPTION:
In a multi-center pragmatic clinical trial, COVID-19 positive patients admitted to 6 United States medical centers were enrolled between March 10 and June 4, 2020. A machine learning algorithm was used to determine which patients were suitable for treatment with hydroxychloroquine.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to covered ward and tested positive for COVID-19
* Patient had COViage applied to electronic health record data within four hours of COVID-19 test

Exclusion Criteria:

* Patient not admitted to covered ward or tested negative for COVID-19
* Patient had COViage applied to electronic health record data greater than four hours after COVID-19 test

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2020-06-04 (Actual)

PRIMARY OUTCOMES:
Mortality outcome | Through study completion, an average of 3 months
  Time to in-hospital death

CONTACTS AND LOCATIONS:
Locations (1):
- Dascena, Oakland, California, United States